CLINICAL TRIAL: NCT01889082
Title: Recruiting and Retaining Young Adults in Behavioral Weight Loss Treatment
Acronym: SPARKRVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM14857; 5K23DK083440-06 (NIH)
Record Dates: First submitted 2013-03-11; First posted 2013-06-28 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: Obesity; weight loss; young adults
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Face to Face Behavioral Weight Loss (Active Comparator): 12-week treatment program consisting of weekly, in-person group meetings and brief, bi-weekly individual check-ins
  Interventions: Behavioral: Behavioral Weight Loss Intervention for Young Adults
- Web Based Behavioral Weight Loss (Active Comparator): 12-week treatment program consisting of an initial in-person group session (weight loss 101 and intro to website), followed by weekly web-based program and e-coaching
  Interventions: Behavioral: Behavioral Weight Loss Intervention for Young Adults
- Web Based Behavioral Weight Loss Plus Optional Group Sessions (Active Comparator): 12-week treatment program consisting of an initial in-person group session (weight loss 101 and intro to website), followed by weekly web-based program and e-coaching. Participants in this arm will also have the option to attend several experiential group sessions that will help those interested to apply the material and skills they are being taught (e.g., cooking demonstration, circuit training). *New material / content is not provided in these optional sessions, rather they are meant to serve as a place to practice applying the core content from the lessons.
  Interventions: Behavioral: Behavioral Weight Loss Intervention for Young Adults

INTERVENTIONS:
Behavioral: Behavioral Weight Loss Intervention for Young Adults

SUMMARY:
A randomized pilot study will be conducted, the goal of which is to determine which format represents the most viable approach to behavioral weight loss treatment with 18-25 year olds. Specifically, participants will be randomized to one of three arms; all arms will receive a 12-week behavioral weight loss intervention, including identical dietary, physical activity, and weight loss prescriptions.

DETAILED DESCRIPTION:
A randomized pilot study will be conducted, the goal of which is to determine which format represents the most viable approach to behavioral weight loss treatment with 18-25 year olds. Specifically, participants will be randomized to one of three arms; all arms will receive a 12-week behavioral weight loss intervention, including identical dietary, physical activity, and weight loss prescriptions. Behavioral goals / prescriptions will be the same, and basic content delivered will also be the same; only the format by which the intervention is delivered will differ among the treatment arms. A total of 45-55 participants, 18-25 years of age, with a BMI between 25 and 45 kg/m2 will be randomized to one of three groups: 1) Face-to-face brief behavioral weight loss (FBWL), 2) Web-based brief behavioral weight loss (WBWL), or 3) Web-based brief behavioral weight loss PLUS optional group sessions (WBWL Plus). Assessments will take place at 0 (baseline), 3 (post-treatment), and 6 months (follow-up).

ELIGIBILITY:
Inclusion Criteria: Between 18-25 years of age. Body Mass Index (BMI) between 25 and 45 kg/m2. Men and women will be recruited. All race and ethnic groups will be recruited.

-

Exclusion Criteria:

1. Currently receiving treatment for Type 2 Diabetes, hypertension, hyperlipidemia, or report a history of cardiovascular disease.
2. Other health problems which may influence the ability to walk for physical activity or be associated with unintentional weight change, including cancer treatment within the past 5 years or tuberculosis.
3. Report a history of, or current diagnosed DSM-IV-TR eating disorder (i.e., anorexia nervosa or bulimia nervosa) or any current compensatory behaviors (e.g., vomiting, laxative use, excessive exercise).
4. Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
5. Report a history of any psychotic disorder, bipolar disorder, or organic brain syndromes; report hospitalization for any psychiatric disorder within the last 12 months.
6. Are currently participating in a weight loss program and/or taking weight loss medication.
7. Lost > 5% of body weight during the past 6 months or history of bariatric surgery.
8. Participation in any other research study that may interfere with this study.
9. Intend to move outside of the surrounding area within the time frame of the investigation or will be out of town / unavailable for three or more weeks during the initial intervention period.
10. Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation.
11. Failure to complete screening appointments.

    -

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Adherence and Retention | 12 Weeks
  Primary Aims Include:
  1. To determine whether it is feasible to engage and retain 18-25 year olds in a clinic-based, face-to-face BWL program, as evidenced by achieving >80% attendance at sessions and >80% retention at post-treatment assessment visits.
  2. To determine whether it is feasible to engage and retain 18-25 year-olds in a web-based BWL program, as evidenced by achieving >80% completion of reporting activities and >80% retention at post-treatment assessment visits.
  3. To determine whether engagement and retention is improved in the web-based BWL program by the addition of optional in-person sessions.

SECONDARY OUTCOMES:
Weight Loss | 3 Months

OTHER OUTCOMES:
Satisfaction and Acceptability | 3 Months
  We will assess satisfaction, perceived quality of the interventions, perceived relevance for young adults. Satisfaction will be measured on a likert scale. Acceptability will be measured by engagment.
Waist Circumference | 3 Months
Body Composition | 3 Months
Blood Pressure | 3 Months
Dietary Behaviors | 3 Months
Physical Activity | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G LaRose, PhD, Principal Investigator — Virginia Commonwealthy University
Locations (1):
- Virginia Commonwealth University School of Medicine, Richmond, Virginia, United States

REFERENCES:
- [Derived] LaRose JG, Tate DF, Lanoye A, Fava JL, Jelalian E, Blumenthal M, Caccavale LJ, Wing RR. Adapting evidence-based behavioral weight loss programs for emerging adults: A pilot randomized controlled trial. J Health Psychol. 2019 Jun;24(7):870-887. doi: 10.1177/1359105316688951. Epub 2017 Jan 29. PMID 28810394